CLINICAL TRIAL: NCT06533176
Title: Towards Real-time Personalized Brain State-dependent TMS to Enhance Poststroke Hand Rehabilitation
Brief Title: Real-time Personalized Brain State-dependent TMS After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Hussain (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Sara Hussain, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 202504299; R03HD114188 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain state-dependent TMS during strong states (Experimental)
  Interventions: Device: Personalized brain state-dependent single-pulse TMS
- Brain state-dependent TMS during random states (Active Comparator)
  Interventions: Device: Personalized brain state-dependent single-pulse TMS

INTERVENTIONS:
Device: Personalized brain state-dependent single-pulse TMS — Single-pulse TMS will be applied to the lesioned hemisphere during brain activity patterns associated with strong residual corticospinal tract activation and random brain activity patterns.

SUMMARY:
Transcranial magnetic stimulation (TMS) interventions could feasibly strengthen residual corticospinal tract (CST) connections and enhance recovery of paretic upper extremity function after stroke. This project will test whether personalized brain state-dependent TMS can activate the residual corticospinal tract better than standard TMS, and evaluate the relationship between this activation and upper extremity motor impairment.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) interventions could feasibly strengthen residual corticospinal connections and enhance recovery of paretic upper extremity function after stroke. To maximize the therapeutic effects of such interventions, they must be delivered during poststroke brain activity patterns during which TMS best activates the residual corticospinal tract and enhances neural transmission within it (i.e., brain state-dependent TMS). In this study, the investigators will test the feasibility of real-time, personalized brain state-dependent TMS in chronic stroke survivors. The investigators will also quantify the relationship between personalized poststroke brain state-dependent activation of the residual corticospinal tract and upper extremity motor impairment; results will inform future clinical trial inclusion criteria.

Participants will visit the laboratory for two days of testing that are separated by at least one night of sleep. On Day 1, participants will provide their informed consent. The MacArthur Competence Assessment Tool and the Frenchay Aphasia Screening Test will be used to evaluate consent capacity and confirm the presence of expressive aphasia as needed. Afterwards, the investigators will complete eligibility screening and clinical assessment of upper extremity motor impairment using the Upper Extremity Fugl-Meyer Assessment, measurements of grip and pinch strength, and a dexterity measurement that requires participants to place small pegs into round holes. Participants will then be screened for the presence of residual corticospinal connections from the lesioned hemisphere to an affected upper extremity muscle at rest. Recording electrodes will be attached to multiple affected arm muscles in order to record TMS-evoked twitches in these muscles. During this screening procedure, single-pulse TMS will be applied to each point of a 1 cm resolution grid covering primary and secondary motor areas of the lesioned hemisphere at maximum stimulator output. If TMS reliably elicits a muscle twitch in any of the recorded muscles, that participant will be considered to have residual corticospinal connections and will be eligible for the full study. If no muscle twitch can be elicited in any of these muscles, that participant will not be eligible for the full study. Afterwards, all recording electrodes will be removed and the participant will leave the laboratory.

On Day 2, participants will return to the laboratory. The investigators will place recording electrodes on the scalp using a swim-type cap. The investigators will also place recording electrodes on the most distal affected arm muscle in which a twitch was most reliably observed during Day 1 as well as four additional muscles of the affected arm. After determining the location at which TMS best elicits muscle twitches, the investigators will determine the lowest possible intensity at which TMS elicits muscle twitches at least half of the time. Then, they will deliver 6 blocks of 100 single TMS pulses while the participant rests quietly with their eyes open; stimulation will be delivered at an intensity that is 20% greater than the lowest possible intensity at which TMS elicits muscle twitches at least half of the time. Afterwards, the investigators will use the muscle and brain activity recordings acquired during these 6 blocks to build a personalized mathematical model that identifies which patterns of brain activity correspond to the largest TMS-evoked muscle twitches. The investigators will then use this model to detect the occurrence of these brain activity patterns in real-time; when these patterns are detected, single TMS pulses will be delivered. For comparison, the investigators will also deliver single TMS pulses during random brain activity patterns. Afterwards, all recording electrodes will be removed, participation will be complete, and the participant will leave the laboratory.

The investigators will recruit a total of 37 chronic stroke survivors for this study. The number of participants needed for this study was determined from their preliminary studies and previous studies that explored the relationship between variability in corticospinal tract activation (a necessary component of building robust personalized mathematical models) and corticospinal tract integrity (a correlate of motor impairment and recovery potential).

ELIGIBILITY:
-Presence of residual upper extremity hemiparesis, defined as any of the following: Fugl Meyer Upper Extremity Score <66, Wolf Motor Function Test Score <70, Affected hand performance on the 9-Hole Peg Test >= 10% worse than unaffected hand, Affected hand pinch, key, or power grip performance >= 10% worse than unaffected hand,

* Occurrence of ischemic or hemorrhagic stroke >= 6 months before participation
* Mini Mental State Exam score > 24
* Willingness and ability to provide informed consent
* No history of neurological disease and/or neurological injury other than stroke
* No TMS contraindications, including but not limited to:

Cardiac pacemaker, Cochlear implant, Cortical stimulator, Deep brain stimulator, Vagus nerve stimulator, Cervical spine epidural stimulation, Ventriculoperitoneal shunt, Ferromagnetic metallic implants above the level of the seventh cervical vertebra, Seizure in the last 12 months while taking anti-epilepsy medication, History of adverse reactions to TMS or peripheral nerve stimulation, Current, suspected, or planned pregnancy, Any recent changes (within the last month) to medication use

- Presence of residual corticospinal connections innervating an affected upper extremity muscle following stimulation of the lesioned hemisphere (i.e., MEP+), evaluated at rest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
MEP amplitudes | 1 week
  Peak-to-peak MEP amplitudes elicited by single TMS pulses delivered during personalized brain activity patterns corresponding to strong corticospinal transmission and random brain activity patterns will be measured. At the individual participant level, all MEP amplitudes will be normalized to the mean MEP amplitude observed in that participant. Mean normalized MEP amplitudes will be used to calculate the percentage MEP amplitude difference between the two brain activity patterns (i.e., strong and random).
Upper Extremity Fugl-Meyer Assessment Scores | 1 week
  Scores obtained for each participant during the Upper Extremity Fugl-Meyer Assessment will be calculated. This will provide a single impairment score that will be correlated with the percentage MEP amplitude difference between brain activity patterns reflecting strong corticospinal transmission and random brain activity patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States